CLINICAL TRIAL: NCT06313619
Title: Decreasing Irrational Antimicrobial Use in Bangladesh: A Digital Intervention Program
Acronym: SmartAMR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Md Atiqul Haque, Professor, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BSMMU/20236831
Record Dates: First submitted 2023-11-25; First posted 2024-03-15 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Resistance Bacterial; Increased Drug Resistance; Drug Resistance, Microbial
Keywords: Anti-microbial resistance; Digital intervention; Irrational use

STUDY DESIGN:
Intervention Model Description: A single group of pharmacy drug sellers were trained on using a digital pharmacy management system including record keeping, AI symptom checker, telemedicine services, counselling, and SMS reminder for dose completion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Digital Pharmacy Intervention (Experimental): A total of 39 pharmacy will be included in the intervention. The digital intervention named "SmartAMR" will be introduced among them. The participants will install the mobile app and use it to keep record of the antimicrobial sales in a central database.
  Interventions: Combination Product: SmartAMR

INTERVENTIONS:
Combination Product: SmartAMR — "SmartAMR" is a digital system including a mobile app that helps keeping record of medicine sales, sending auto-generated messages to the consumers to remind them about medicine taking time and completing doses. It also poses a symptom checker driven by artificial intelligence and a telemedicine service.

SUMMARY:
We developed 'SmartAMR', a digital pharmacy system featuring real-time records, symptom checks, telemedicine, counselling, and medication reminders. This study aims to assess its feasibility, acceptability, and effectiveness within community pharmacy settings in Bangladesh.

A before-after designed pilot quasi experimental study will be conducted in urban areas. Data will be collected in both qualitative and quantitative methods. Multi-cluster sampling method will be used to select study locations. Pharmacists or drug sellers and patients aged more than 18 years and located within selected intervention areas will be our target population. A baseline survey will be conducted among the pharmacy volunteers to evaluate their knowledge, perception, and practice of rational use of anti-microbials prior to any intervention. Additionally, a household survey will be conducted among community members applying systematic random sampling where one adult from every selected household will be approached maintaining gender equality. After collecting the baseline data, intervention will be given to the community people through awareness building campaign and distributing leaflets and posters on rational use of anti-microbials. After three months, a follow-up survey will be conducted with the same questionnaire. For quantitative portion of the study, all the medicine shops in the selected study areas will be included in the study sample. For qualitative part, the sample will be selected purposively until data saturation and a total of 8 experts will be interviewed. Two sets of questionnaires for pharmacy volunteers and the community dwellers will be prepared based on literature review that will include health literacy questions regarding anti-microbial use. The questionnaire for the follow-up data collection will include some additional questions regarding effectiveness, acceptability, adoption, feasibility, and cost of the intervention.

DETAILED DESCRIPTION:
The misuse, irrational, or overuse of antibiotics, antibiotic/antimicrobial resistance (AMR) is a global threat to human health. Even though the awareness of the potential threat from AMR is widespread, studies and monitoring programs describing the present situation are lacking. The presence of a 'pluralistic' health system and a large informal sector involving unqualified drug dispenser/providers/practitioners in Bangladesh is a matter of grave concern for the rising antimicrobial resistance situation in the country. An estimated 63% of antibiotic prescriptions are from unqualified providers. Besides, misconception about antibiotics is very common in Bangladesh. Meanwhile, the use of antibiotics in animal food production with insufficient veterinary supervision for therapeutic purposes which poses the risk of antimicrobial resistance transmission in the food chain. Without adherence to national regulations, unnecessary and inappropriate prescriptions become common practice, particularly in rural areas. Domestic drug industries contribute to easily accessible and affordable drugs. To tackle this problem, prescriptions and sales of antibiotics need to be regulated and integrated in a national HMIS. Awareness programs for antibiotic providers that promote understanding of antibiotics and antibiotic resistance through tailored interventions may be helpful in changing current antibiotic sales practices. Therefore, this study will attempt to identify the underlying causes of irrational anti-microbial usage in Bangladesh, which were grouped into four interlinked areas - lack of awareness among patients/ consumers (demand side), perverse incentives and lack of knowledge among providers (supply side), poorly regulated pharmaceutical marketing and retail sales (regulatory side) and lack of data and research evidence to support awareness raising and policymaking (enabler).

This is a pioneering study in Bangladesh that introduces a comprehensive digital pharmacy management system, demonstrating its feasibility and acceptability while highlighting potential challenges. The intervention showed promise in improving record-keeping, raising awareness, and promoting rational antibiotic use. The cloud-based server of this system allows its integration with existing government data systems, providing it the privilege to scale up to a nationwide level and achieve sustainability. With adequate support and strategies to mitigate profit-driven noncompliance, such pharmacy-based interventions can play a vital role in national efforts to combat AMR.

The study is expected to bring light upon a comprehensive understanding of the current level of knowledge, perception and practice of irrational use of anti-microbials among target population. Furthermore, a digital intervention design will be produced and piloted to reduce irrational use of anti-microbials after considering its effectiveness. The wide range of the study findings will aid in assessing the acceptability, adoption, feasibility and cost of the intervention to make recommendations on sustainability and scaling up of the intervention programs.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and above
* Registered drug seller/pharmacist
* Permanent residents of the study areas
* Willing to participate

Exclusion Criteria:

* Disoriented or critically ill

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2023-10-23 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Irrational usage of anti-microbials | 12 weeks
  Irrational usage of anti-microbials was demonstrated by number and pattern of purchasing of anti-microbials
Acceptance rate | 12 weeks
  Number of pharmacy agreed and accepted the intervention and install the mobile app.
Completion rate | 12 weeks
  The number of pharmacy who use the mobile app for the total duration of intervention.
AMR Knowledge | Before and 12 weeks after the intervention
  Change in knowledge about antimicrobial resistance among the participants was assessed using a knowledge scale "AMR knowledge scale" that contained 31 questions. The score range will be 0 to 31, with greater score representing better knowledge.
AMR attitude | Before and 12 weeks after the intervention
  Participants' attitude towards antimicrobial resistance was evaluated by a three-point Likert-type scale "AMR attitude scale", containing 14 attitude statements. The score range will be 14 to 42, with greater score representing better knowledge.
AMR practice | Before and 12 weeks after the intervention
  Participants' practice regarding irrational antimicrobial usage is assessed by a practice scale "AMR practice scale", containing 9 items. Answers to the practice questions are taken on a rating scale (0=never; 1 = rarely; 2 = sometimes; 3 = frequently). Practice score ranges from 0 to 27. Higher score indicates better practice.

CONTACTS AND LOCATIONS:
Overall Officials: M Atiqul Haque, PhD, Study Director — Bangladesh Medical University
Locations (1):
- Bangladesh Medical University, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No